CLINICAL TRIAL: NCT06054022
Title: Comparing Intraoperative High Flow Nasal Cannula Therapy and Convetional Oxygen Therapy in Preventing Perioperative Hypoxaemia In Elderly Patients Undergoing Orthopaedic Surgery: A Randomized Controlled Study
Brief Title: Usage of High Flow Nasal Cannula in Preventing Desaturations in Elderly Patients Going for Lower Limb Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FFP-2020-245
Record Dates: First submitted 2020-11-10; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hypoxemia During Surgery; Atelectasis
Keywords: high flow nasal cannula; elderly; orthopaedic; hypoxaemia; regional anaesthesia
MeSH Terms: conditions — Pulmonary Atelectasis; Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: there will be no masking except for the radiologist who compares the postoperative chest x-ray with the baseline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient receiving high flow nasal cannula (A) (Experimental): Patient will be put on high flow nasal cannula at a fixed flow of 50L/min, at Fio2 0.3% throughout surgery. Oxygen therapy will be discontinued once surgery ends. FiO2 will be titrated by 0.1 increment to a SpO2 of ≥94%.
  Interventions: Device: high flow nasal cannula
- patient receiving nasoprong oxygen 2 L/min (Active Comparator): Patient will be put nasoprong oxygen 2L/min throughout surgery. Oxygen therapy will be discontinued once surgery ends. FiO2 will be titrated by 0.1 increment to a SpO2 of ≥94%.
  Interventions: Device: nasoprong oxyen 2Litres per minute

INTERVENTIONS:
Device: high flow nasal cannula — high flow nasal cannula provides heated and humidified gas to the airways via nasal prongs at a prescribed accurate fraction of inspired oxygen (FiO2) ranging from 0.21 to 1.0 and with a higher flow rate of up to 60 litres per minute
  Arms: patient receiving high flow nasal cannula (A)
Device: nasoprong oxyen 2Litres per minute — nasoprong @L/min will deliver approximately a FiO2 of 0.3. subsequently, if incremental O2 is needed, patient will be provided with ventimask 40% and so forth
  Arms: patient receiving nasoprong oxygen 2 L/min

SUMMARY:
To study the effect of high flow nasal cannula in comparisons with nasoprong used intraoperatively in patients oxygenation status

DETAILED DESCRIPTION:
To observe the effect of high flow nasal cannula used intraoperatively compared to normal oxygen therapy (nasoprong) at a same fraction of inspired oxygen (FiO2) in elderly patients who are going for orthopaedic surgeries under central neuraxial block.

oxygenation will be access with intermittent blood gas. atelectasis will be access via chest x-ray , compared to a baseline chest x-ray, validated by a blinded radiologist

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) I, II or III patients.
2. Patients age 60 years and above
3. Patients scheduled for total knee replacement therapy and hip surgeries under central neuraxial block under the elective and emergency list.

Exclusion Criteria:

1. Patients with pre-operative spO2<94%
2. Patients delirious or demented / unable to give consent.
3. Patients with pre-existing pneumonia (defined as the initiation of antibiotics for suspected infection with one or more of the following: new or changed sputum; new or changed lung opacities; fever; white blood cell count >12 × 109 litre-1 )15
4. BMI ≥35

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incident of intraoperative desaturation | From induction time until end of surgery
  desaturation is taken as any spO2 <94%
Patient comfort on high flow nasal cannula | At end of surgery till discharge to ward (recovery area)
  Patient rate comfort level using Visual Numerical Scale. The scale of 1 to 5 with 1 being extreme discomfort, 3 neutral and 5 extreme comfort
Atelactasis | From end of operation until 24 hours post surgery
  Incident of postoperative atelectasis by compraring the preoperative and postoperative chest x ray by a radiologist

SECONDARY OUTCOMES:
Length of hospital stay | Time of hospital admission to time of discharge up to 30 days which ever come first
  Duration of hospital admission from the time of patient admitted to the hospital, until discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Syarifah noor nazihah binti sayed masri, MD, Principal Investigator — National University of Malaysia
Locations (1):
- Universiti Kebansaan Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No